CLINICAL TRIAL: NCT03246932
Title: The Effectiveness of a Peer-led Psycho-education Group in Schizophrenia: A Multi-site Randomised Controlled Trial
Brief Title: Peer-led Psycho-education for Schizophrenia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Hospital Authority, Hong Kong (Other Government); Jilin University Medical Science Division (Unknown); Taipei Medical University (Other)
Responsible Party: Principal Investigator, Prof. Wai Tong CHIEN, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CWai-Tong
Record Dates: First submitted 2017-08-08; First posted 2017-08-11 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Schizophrenia
Keywords: peer expert or specialist; psycho-education; schizophrenia; outpatients
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blinded to the group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Peer-led psycho-education group (Experimental): A structured, researcher-designed peer expert-led psycho-education program (6 months), comprised of 12 bi-weekly, 2-hour group sessions (10-12 patients per group). The program was based on the psycho-education and self-help, problem-solving programs by Chien et al. (2010) and Lehman et al. (2004).
  Interventions: Behavioral: Peer-led psycho-education group; Other: Routine psychiatric care
- Routine psychiatric care (Other): Routine psychiatric outpatient care, including medication, psychiatric consultation in outpatient clinic, brief education by psychiatric nurses, financial and social welfare advices by social workers, and individual counseling by clinical psychologist.
  Interventions: Other: Routine psychiatric care
- Profession-led psycho-education group (Active Comparator): A psycho-education group program (12 sessions, bi-weekly) based on Dr. Macpherson's Family Psychoeducation Program in 1996 and Chien and Bressington's one in 2014/15 will be used.
  Interventions: Behavioral: Profession-led psycho-education group; Other: Routine psychiatric care

INTERVENTIONS:
Behavioral: Peer-led psycho-education group — A structured, researcher-designed peer-led psycho-education program (6 months), comprising of 12 bi-weekly, 2-hour group sessions.
  Arms: Peer-led psycho-education group
Behavioral: Profession-led psycho-education group — A psychoeducation group program (12 sessions, bi-weekly).
  Arms: Profession-led psycho-education group
Other: Routine psychiatric care — Routine psychiatric outpatient care, or Treatment-as-usual (TAU).

SUMMARY:
Profession-led psycho-education programs for people with schizophrenia are evidenced to improve patients' knowledge about the illness, mental state and relapse rate. Nevertheless, other benefits to patients, for example, their functioning and insight into illness or to be substantive in a longer term (>12 months) are inconsistent and uncertain, especially in Asian populations. This single-blind multi-site randomized clinical trial was to test the effects of a peer-expert-led psycho-education group intervention (in addition to usual care) for adult patients with schizophrenia spectrum disorders over a 24-month follow-up, in comparison to a profession-led psycho-education group or treatment-as-usual only.

DETAILED DESCRIPTION:
Objectives: This study is to test the effectiveness of a peer-expert-led psycho-education group programme for Chinese outpatients with schizophrenia spectrum disorders over an 24-month follow-up. The program is an integrated,psycho-education program that addresses patients' knowledge and self-management of schizophrenia and problem-solving skills. Methods: A single-blind, multi-site randomized controlled trial will be conducted with 342 Chinese patients with schizophrenia in Hong Kong, China and Taiwan. In each of three study sites, the participants will be randomly selected from the eligible patient list (i.e., 114 subjects from each study site) and after baseline measurement, be assigned to either the peer-led psycho-education program, profession-led psycho-education group, or usual psychiatric care. The patients' mental and psychosocial functioning, insights into illness, and their re-hospitalization rates will be measured at recruitment and at one week, and 6, 12 and 24 months after completing the interventions. Hypothesis: The patients in the peer-led psycho-education program will report significantly greater improvements in their symptoms and re-hospitalisation rates (primary outcomes) and other secondary outcomes (e.g., insight into illness and functioning) over the 24-month follow-up, when compared with those in profession-led psycho-education group and/or usual care. Conclusions: The findings will provide evidence whether the peer-led psycho-education group program can better improve Chinese schizophrenia sufferers' psychosocial functioning and reduce their illness relapse.

ELIGIBILITY:
Inclusion Criteria:

* patients, aged 18+, attending one psychiatric outpatient clinic under study;
* diagnosed as schizophrenia and its subtypes according to the Diagnostic and Statistical Manual, 4th Text-Revised Edition, as ascertained by the Structured Clinical Interview (SCID-I);
* having onset of the illness for not >5 years; and
* able to communicate in Cantonese language.

Exclusion Criteria:

* mentally unstable and unfit for study participation at recruitment;
* with co-morbidity of other severe mental health problems such as depression and substance misuse; and
* have recently received or are receiving any structured psychosocial intervention.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 342 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale | from recruitment to 24-month follow-up
  The Positive and Negative Syndrome Scale assesses the severity of psychotic symptoms on three subscales: positive symptoms (7 items), negative symptoms (7 items) and general psychopathology (16 items). will be assessed at recruitment and one week, 6 months, 12 months and 24 months after the interventions completed.
Specific Level of Functioning Scale | from recruitment to 24-month follow-up
  Patients' levels of psychosocial functioning will be assessed with the Specific Level of Functioning Scale at baseline and one week, 6 months, 12 months and 24 months follow-up.

SECONDARY OUTCOMES:
Re-hospitalization rate | from recruitment to 24-month follow-up
  Average amount (number) and length of hospital stay of the patients over previous six months will be assessed at recruitment and one week, 6 months, 12 months and 24 months after the interventions completed.
Six-item Social Support Questionnaire | from recruitment to 24-month follow-up
  Patients' perceived social support will be assessed with the Six-item Social Support Questionnaire at baseline and one week, 6 months, 12 months and 24 months follow-up.

OTHER OUTCOMES:
Insights to illness and treatment | from recruitment to 24-month follow-up
  Patients' insight and attitudes to illness and treatment will be measured with the Insight and Treatment Attitudes Questionnaire at recruitment and one week, 6 months, 12 months and 24 months after the interventions completed.

CONTACTS AND LOCATIONS:
Overall Officials: WT Chien, PhD, Principal Investigator — CUHK
Locations (2):
- Jilin Medical College, Jilin, Jilin, China
- TM Psy Centre, Tuenmen, NT, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chien WT, Norman I. The effectiveness and active ingredients of mutual support groups for family caregivers of people with psychotic disorders: a literature review. Int J Nurs Stud. 2009 Dec;46(12):1604-23. doi: 10.1016/j.ijnurstu.2009.04.003. Epub 2009 May 28. PMID 19481205
- [Background] Chien WT, Leung SF, Yeung FK, Wong WK. Current approaches to treatments for schizophrenia spectrum disorders, part II: psychosocial interventions and patient-focused perspectives in psychiatric care. Neuropsychiatr Dis Treat. 2013;9:1463-81. doi: 10.2147/NDT.S49263. Epub 2013 Sep 25. PMID 24109184
- [Background] Chien WT, Clifton AV, Zhao S, Lui S. Peer support for people with schizophrenia or other serious mental illness. Cochrane Database Syst Rev. 2019 Apr 4;4(4):CD010880. doi: 10.1002/14651858.CD010880.pub2. PMID 30946482
- [Background] Chien WT, Bressington D. A randomized controlled clinical trial of a nurse-led structured psychosocial intervention program for people with first-onset mental illness in psychiatric outpatient clinics. Psychiatry Res. 2015 Sep 30;229(1-2):277-86. doi: 10.1016/j.psychres.2015.07.012. Epub 2015 Jul 10. PMID 26193827